CLINICAL TRIAL: NCT04423289
Title: COVID Follow-App: Telematic Monitoring Through a Mobile Application of Patients With COVID-19: A Randomized Clinical Trial
Brief Title: Telematic Monitoring Through a Mobile Application of Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR(AG)182-2020
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Face-to-face Reconsultation to Emergency Room

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Farmalarm (Experimental): Farmalarm app for the follow-up
  Interventions: Other: Farmalarm
- Control (No Intervention): Regular primary care follow-up

INTERVENTIONS:
Other: Farmalarm — Monitoring after COVID-19 discharge from hospital via Farmalarm app
  Arms: Farmalarm

SUMMARY:
Open-label randomized clinical trial, one center, to compare the need for face-to-face re-consultation after discharge for COVID-19 between a telematic monitoring through a mobile app and the regular primary care setting.

DETAILED DESCRIPTION:
A randomized, open-label clinical trial, at one center, a 1100-bed academic hospital, Vall d'Hebron Hospital Universitari, in Barcelona, Spain. Patients who met the enrolment criteria were randomly assigned, in a 1:1 ratio, to be followed by the Farmalarm app or the primary care setting.

Farmalarm is an app for smartphones designed to increase stroke awareness and treatment compliance through visual and audible alerts. The application's software offers versatility to modify the parameters to be monitored and the information to be sent, which were adapted to our purpose.

Intervention was started after the patient was discharged and underwent randomization. At this moment, patients assigned to the study group were given a personal access code ensuring data privacy, and they were lent an intelligent pulse oximeter (SMART PULSE OXIMETER OL-750, LifeVit, Guangdong Biolight Meditech CO., LTD, China). In a 15 minutes interview they were trained in the use of the app, the use of the pulse oximeter and the measurement of some vital signs.

On that same day, the healthcare professional uploaded and scheduled on the web-based platform a personalized program for the following 2 weeks.

To maintain close control of respiratory evolution, patients registered at least 2 times a day their heart rate, respiratory rate, temperature and peripheral capillary oxygen saturation. The intelligent pulse oximeter allowed data to be downloaded directly to the WP every time the patient used it. They also had to answer a symptom survey every day for the same period. The WP allows scheduling alarms and so, in case one of the vital signs or survey responses were altered, the healthcare in charge automatically received a notification, being able to contact immediately the patient. A private chat between the patient and the healthcare responsible for WP was attended every day from 8 AM to 5 PM to answer any doubt.

Patients assigned to control group received regular follow-up at the Primary Care, which used phone calls to monitor patients' symptoms. Depending on the availability of human resources of each Primary Care Centre and the care pressure of the moment, these phone calls were made every 2 days, weekly, or just once during the whole follow-up period.

All patients were followed for two weeks. At the end of follow-up, all patients answered an end-of-follow-up questionnaire and a Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire about global health. The end-of-follow-up interview of experimental group patients was carried by videoconference through the app. Control group patients were telephonically contacted. All patients also answered a Hospital Anxiety and Depression Scale (HADS) the same day of discharge and again at the end of follow-up. 12

ELIGIBILITY:
Inclusion Criteria:

* an age of 18 years or older,
* availability of a mobile device such a phone or a tablet with connectivity to the internet, and
* discharged from hospital after admission for COVID-19 diagnosed by RT-PCR.

Exclusion Criteria:

* health personnel (medical or nursing staff) or
* discharged to care centers or medicalized hotels enabled to complete the period of isolation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Re-consultation | 2 weeks
  Number of patients needing face-to-face re-consultations

SECONDARY OUTCOMES:
Telephone calls | 2 weeks
  Number of patients making telephone calls to emergency services

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Len, MD, PhD, Principal Investigator — Vall d'Hebron Hospital Universitari
Locations (1):
- Vall d'Hebron Hospital Universitari, Barcelona, Spain